CLINICAL TRIAL: NCT04449783
Title: A Cohort Study to Assess the Effectiveness of Preoperative Shielding and N/T RT-PCR Swabbing for Elective Cancer Surgery Patients in the COVID-19 Pandemic
Brief Title: Preoperative Shielding and N/T RT-PCR Swabbing for Elective Cancer Surgery
Acronym: CHICANE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: SP0355
Record Dates: First submitted 2020-06-23; First posted 2020-06-29 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-06

CONDITIONS: Covid19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study patients: Patients undergoing elective cancer surgery, who will receive pre-operative screening including reporting symptoms and nose and throat swabbing 48 hours prior to surgery
  Interventions: Other: pre-operative screening; Other: telephone consult

INTERVENTIONS:
Other: pre-operative screening — reported symptoms plus nose and throat swabbing 48 hrs prior to surgery
Other: telephone consult — telephone consult 14 days (+/- 2 days) to assess for any COVID-19 symptoms

SUMMARY:
trial to assess the effectiveness of pre-operative screening for COVID-19 in patients undergoing elective cancer surgery.

DETAILED DESCRIPTION:
1. Background:

   The optimal method of screening patients for COVID infection before elective cancer surgery is unclear. Provisional data from the international COVIDsurg audit as well as a similar study from China has shown mortality rates of in excess of 20% for COVID +ve patients undergoing surgery and so ensuring patients do not have infection before surgery is critical (1).

   Current practice for the preoperative screening of elective surgical patients involves a period of self-isolation, assessment of self-reported symptoms and nose and throat swab testing. Many patients are asymptomatic with COVID and the false negative rate of RT-PCR nose and throat swabs may be as high as 30% (2,3). Furthermore, we do not know how effective our strategy is at preventing hospital acquired COVID in the days after surgery. Patients are currently going to designated clean (silver) wards postoperatively to reduce this risk with other patient who have tested negatively to the above screening process too
2. Rationale:

The aim of this study is to assess the rate of perioperative COVID in elective surgical patients, and to assess whether RT-PCR swabbing adds any additional value i.e. does it detect clinically important asymptomatic patients.

If asymptomatic patients are diagnosed preoperatively this will reduce perioperative morbidity and mortality as well as confirming this as an appropriate preoperative screening process. Alternatively, should nose and throat swabbing not improve the diagnosis of COVID-19 in asymptomatic patients this trial may stop unnecessary visit to the hospital where they may be more likely to contract COVID-19 and reduce the use of a limited resource.

ELIGIBILITY:
Inclusion Criteria:

* participants capable of giving informed consent,
* gender: Male and Female
* Age: 18 years and above
* Preoperative cancer patients (elective)
* Willing to be contacted by phone after hospital discharge
* Patients listed for inpatient admission postoperatively (cancer patients)

Exclusion Criteria:

* Cancer patients who require non-cancer surgery
* emergency cancer operations
* Patients under the age of 18
* Patients who do not have capacity to consent
* Cancer patients not requiring an inpatient stay postoperatively
* Patients who it was not anticipated would require an inpatient stay preoperatively but required admission after surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients undergoing elective cancer surgery with an inpatient stay
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-08-25 (Estimated); Study Completion 2020-09-25 (Estimated)

PRIMARY OUTCOMES:
diagnosis of COVID before surgery | prior to surgery
  Diagnosis of COVID on day of surgery (based on Clinical symptoms +/- positive swab diagnosis)

SECONDARY OUTCOMES:
diagnosis of COVID after surgery | 14 days post op
  Diagnosis by day 14 (+/-2) post-surgery (based on Clinical symptoms from inpatient notes or telephone consultation +/- positive swab diagnosis)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jones, MBChB, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No
will not be shared